CLINICAL TRIAL: NCT07339462
Title: Feasibility and Acceptability of Critical Time Intervention to Support People With Severe Mental Illness Following Post-acute Hospital Discharge in South Africa
Brief Title: Feasibility and Acceptability of an Intervention to Support People With Severe Mental Illness in South Africa
Acronym: MhINT Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Columbia University (Other); Universiteit Antwerpen (Other); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R34MH131233-01 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Mental Disorders, Severe
Keywords: Severe mental illness; Community-based care; Family empowerment; Recovery; Hospital readmission; Deinstitutionalization; Integrated care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Co-developed health system strengthening intervention (MhINT Recovery)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention arm will be exposed to the following interventions:
  1. A revised referral pathway across tertiary, secondary and primary levels of care, integrated with existing policies;
  2. A psychosocial rehabilitation programme, including a manual and training and mentorship package, introduced to multidisciplinary teams and nursing staff in specialist, regional and district hospitals
  3. A psychosocial rehabilitation programme, including a manual and training and mentorship package, introduced to registered counsellors in PHC facilities
  4. Refresher training on management of severe mental health conditions for physicians and nurses in PHC facilities
  5. A community mental health education and detection toolkit and associated training package for community health worker outreach teams
  6. The Household Champion programme, a psychoeducation, empowerment and support programme to improve caregiver capacity and improve community resource linkages.
  Interventions: Behavioral: Multilevel psychosocial support for people living with severe mental illness and their caregivers
- Control Arm (No Intervention): Service users discharged from acute psychiatric hospitalization to households in the community receiving standard care (i.e. monthly procurement of medicines at the primary healthcare clinic), as well as exposure to improved referral pathways as well as psychosocial rehabilitation on hospital level.

INTERVENTIONS:
Behavioral: Multilevel psychosocial support for people living with severe mental illness and their caregivers — The intervention is the product of a human-centred design process, involving a range of health system actors. The intervention entails 1) A revised, integrated referral pathway across tertiary, secondary and primary levels of care; 2) A psychosocial rehabilitation programme, introduced to multidisciplinary teams and nursing staff in specialist, regional and district hospitals; 3) A psychosocial rehabilitation programme, introduced to registered counsellors in PHC facilities; 4) Refresher training on management of severe mental health conditions for physicians and nurses in PHC facilities; 5) A community mental health education and detection toolkit and associated training package for community health worker outreach teams; 6) The Household Champion programme, a psychoeducation, empowerment and support programme to improve caregiver capacity for care.
  Arms: Intervention Arm

SUMMARY:
Despite commendable progress in developing mental health systems in low-and-middle income countries, critical gaps remain, particularly the development of community-based systems of support for people living with severe mental illness (SMIs). This application will pilot a co-developed health system strengthening intervention programme in a South African district in order to determine its feasibility, appropriateness and limited efficacy in reducing readmission following discharge from acute psychiatric hospitalization. By generating preliminary data on the real-world implementation of a co-developed programme in low-resource contexts in South Africa, this application seeks to build on an existing foundation of research partnerships and local government collaboration to develop a transitional support intervention that could yield significant and tangible impacts on people living with SMIs in low-resource communities.

DETAILED DESCRIPTION:
The development of appropriate and effective community-based care for people living with severe mental illness (SMIs) continues to be a global challenge, especially in low-and-middle income countries (LMICs). A particularly damaging cycle emerges when people with SMIs are admitted to hospital for acute psychiatric treatment, discharged back into community settings without appropriate support, only to be readmitted again due to psychiatric relapse. This "revolving door" phenomenon is a multilevel challenge to mental health systems, including in countries such as South Africa, with little to no formal community-based support systems for people living with SMIs. Several innovative strategies have been developed to address hospital re-admission, while co-development approaches such as human-centred intervention development have shown much promise in generating improved outcomes. The proposed research project aims to explore the feasibility and limited efficacy of a co-developed health system strengthening intervention programme in a South African district in order to determine its feasibility, appropriateness and limited efficacy in reducing readmission following discharge from acute psychiatric hospitalization.

Specifically, a multi-level helath system strengthening intervention programme has been co-developed, which include 1) the improvement of referral processes across healthcare facilties; 2) the implementation of a psychosocial rehabilitation programme across tertiary, secondary and primary healthcare facilities; 3) the implementation of clinical guidelines refresher training for clinicials on primary healthcare level; 4) the implementation of a structured outreach programme by community health workers following discharge; and 5) the implementation of a Household Champion programme to empower households for better support at home. This package will be piloted in a parallel arm feasibility trial in the uMgungundlovu District Municipality in KwaZulu-Natal, South Africa. We will train registered councellors to deliver psychosocial rehabilitation on primary healthcare level in tandem with nursing staff, train community health workers to work with existing outreach teams to implement the Community Mental Health Education and Detection programme during routine household visits, and will recruit a training and quality improvement team to coordinate, support and mentor training and improvement for the referral pathway and clinician refresher training. Fourty-three people who have been admitted for acute psychiatric reasons will be recruited for each of the two arms. The intervention arm will receive the full intervention package, while the control arm will receive care as usual as well as improved referral and discharge readiness on hospital level. The primary aim is to determine whether enrollment to the full intervention package will reduce the likelihood of people discharged from acute psychiatric hospitalization after 4 months, compared to those in the control group. Secondary measures include the effects of the intervention on service users (in terms of stigma, medication adherence, and recovery) after 4 months; and qualitative measures of feasibility in terms of the acceptability, demand, implementation, practicality, adaptation, integration, and potential for expansion of the intervention. Taken together, the quantitative and qualitative data will provide an indication of the feasibility and limited efficacy of the co-developed intervention package.

ELIGIBILITY:
Service user inclusion criteria:

* Adults (aged 18 years and above);
* Being admitted to the psychiatric ward of a hospital for observation and treatment due to an acute psychiatric event, based on ICD diagnosis on patient charts according to the following criteria:

  * F20-29 including schizophrenia, delusional disorders, schizotypal disorders, acute polymorph psychotic disorders, schizoaffective disorders
  * F30-39 Mood [affective] disorders with psychoses
  * F30.2 Mania with psychotic symptoms
  * F31.2 Bipolar affective disorder, current episode manic with psychotic symptoms
  * F31.5 Bipolar affective disorder, current episode severe depression with psychotic symptoms
  * F32.3 Severe depressive episode with psychotic symptoms
  * F33.3 Recurrent depressive disorder, current episode severe with psychotic symptoms
* Determined by the attending psychiatrist to be discharged into community settings following appropriate recovery from the psychiatric event;
* Willing and able to participate in the intervention programme
* Resides with a caregiver (which could be a family member or member of the household).
* Resides within the geographic boundaries of uMgungundlovu

Service user exclusion criteria:

* Under 18 years of age
* Are indicated by their chart history to have the following conditions:

  * Active suicidal ideation
  * Substance abuse or dependence as primary diagnosed psychiatric condition
  * Personality disorders
  * Serious cognitive or other sensorial impairment likely to preclude informed consent and reliable assessment
* Does not reside with a caregiver
* Does not reside within the geographic boundaries of uMgungundlovu

Caregiver inclusion criteria

* Adults (aged 18 years and above)
* Willing and able to participate in the intervention programme
* Resides with a caregiver (which could be a family member or member of the household).
* Resides within the geographic boundaries of uMgungundlovu

Caregiver exclusion criteria

* Adults (aged 18 years and above)
* Willing and able to participate in the intervention programme
* Resides with a caregiver (which could be a family member or member of the household).
* Resides within the geographic boundaries of uMgungundlovu

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in rate of hospital psychiatric re-admission among people living with severe mental illness, as assessed by medical records, at 4 months. | From enrollment to 4 months
  The proportion of intervention arm participants who have not relapsed and re-hospitalised for an acute psychiatric event within a period of four months since enrolment, compared to control arm participants, as measured by trial monitoring data.

SECONDARY OUTCOMES:
Change in recovery score among people living with severe mental illness, as assessed by the total score on the Recovery Assessment Scale - Domains and Stages (RAS-DS), at 4 months | Baseline, 4-month follow-up fieldworker-administered questionnaire
  The proportion of intervention arm participants who have shown changes in recovery scores, as measured by the Recovery Assessment Scale - Domains and Stages (RAS-DS), following an acute psychiatric event within a period of four months since enrolment, compared to control arm participants.
  4-point Likert-type scale: Untrue, A bit untrue, A bit true, Completely true
  Hancock N, Scanlan JN, Honey A, Bundy AC, O'Shea K. Recovery Assessment Scale - Domains and Stages (RAS-DS): Its feasibility and outcome measurement capacity. Aust N Z J Psychiatry. 2015 Jul;49(7):624-33. doi: 10.1177/0004867414564084. Epub 2014 Dec 19. PMID: 25526940; PMCID: PMC4941096.
Change in internalized stigma score among people living with severe mental illness, as assessed by the total score on the Brief version of the Internalized Stigma of Mental Illness (ISMI) scale, at 4 months | Baseline, 4-month follow-up fieldworker-administered questionnaire
  The proportion of intervention arm participants who have shown changes in internalized stigma as measured by the Brief version of the Internalized Stigma of Mental Illness (ISMI) scale, following an acute psychiatric event within a period of four months since enrolment, compared to control arm participants.
  4-point Likert-type scale: Strongly disagree, Disagree, Agree, Strongly agree
  Matshabane OP, Appelbaum PS, Faure MC, et al. Lessons learned from the translation of the Internalised Stigma of Mental Illness (ISMI) scale into isiXhosa for use with South African Xhosa people with schizophrenia. Transcultural Psychiatry. 2023;0(0). doi:10.1177/13634615231168461
Change in treatment adherence score among people living with severe mental illness, as assessed by the total score on a tailored scale, at 4 months | Baseline, 4-month follow-up fieldworker-administered questionnaire
  The proportion of intervention arm participants who have shown changes in treatment adherence scores as measures by a tailored measure, following an acute psychiatric event within a period of four months since enrolment, compared to control arm participants.
Description of stakeholder views regarding the acceptability of the MhINT Recovery intervention after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the degree to which the MhINT Recovery intervention is deemed acceptable to people receiving the intervention, their caregivers, healthcare workers, managers, and policymakers, after four months of implementation.
Description of perceptions of stakeholders regarding the demand of the MhINT Recovery intervention after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the degree to which the MhINT Recovery intervention meets the demands of people receiving the intervention, their caregivers, healthcare workers, managers, and policymakers, after four months of implementation.
Description of perceptions of stakeholders regarding the barriers and facilitators of the implementation of MhINT Recovery, in terms of the Consolidated Framework for Implementation Research (CFIR) domains, after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure describing barriers and facilitators in implementation of the MhINT Recovery intervention, in terms of the Consolidated Framework for Implementation Research (CFIR) domains (Inner, Outer, Implementation, Innovation, Individual and Implementation), after four months of implementation.
Description of perceptions of stakeholders regarding the practicality of the MhINT Recovery intervention, after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the degree to which the MhINT Recovery intervention is deemed to be practical by people receiving the intervention, their caregivers, healthcare workers, managers, and policymakers, after four months of implementation.
Description of perceptions of stakeholders regarding the degree to which the MhINT Recovery intervention can be adapted for specific subgroups after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the degree to which the MhINT Recovery intervention can be adapted to the needs of different subgroups of people receiving the intervention, after four months of implementation.
Description of perceptions of stakeholders regarding the degree to which the MhINT Recovery intervention can be integrated into the local health system after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the degree to which the MhINT Recovery intervention is perceived to be integrated with the local health system, after four months of implementation.
Description of perceptions of stakeholders regarding the potential of scaling the MhINT Recovery intervention in future, after 4 months of implementation | From enrollment to the end of the intervention at 4 months
  A qualitative measure of the perceived potential of the MhINT Recovery intervention to be scaled from trial to routine and sustained service changes for people living with severe mental illness, after four months of implementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Msunduzi Local Municipality, Pietermaritzburg, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT07339462/Prot_SAP_ICF_000.pdf